CLINICAL TRIAL: NCT04850729
Title: An Observational Study of Relationship Between Perioperative Treatment Efficacy and The Tumor Microenvironment for Locally Advanced Resectable Gastric and Gastro-oesophageal Junction Adenocarcinoma
Brief Title: Relationship Between Perioperative Treatment Efficacy and The Tumor Microenvironment for Locally Advanced Resectable Gastric Cancer.
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-082
Record Dates: First submitted 2021-04-18; First posted 2021-04-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Cancer; Tumor Microenvironment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
Perioperative drug treatment has gradually become the standard regimen for locally advanced gastric cancer, whereas only a subset of patients could benefit from it. Therefore, one major challenge for perioperative drug treatment is to construct promising biomarkers and to screen out potential beneficial patients. Recent evidence has revealed that tumor microenvironment (TME) is highly associated with the prognosis of gastric cancer. Meanwhile, tumor microenvironment score (TMEscore) established with transcriptomic data is a robust biomarker for predicting prognosis and guiding individualized immunotherapy strategies. However, its predictive value for perioperative drug treatment outcomes warrants further exploration and validation. The study is a multi-center, observational study to evaluate the relationship between the efficacy of perioperative treatment and tumor microenvironment in patients with locally advanced resectable gastric and gastro-oesophageal junction adenocarcinoma, aiming at further determining the predictive value of TMEscore and establishing a comprehensive treatment-efficacy evaluation system for gastric cancer.

DETAILED DESCRIPTION:
Perioperative drug treatment has gradually become the standard regimen for locally advanced gastric cancer, whereas only a subset of patients could benefit from it. Therefore, one major challenge for perioperative drug treatment is to construct promising biomarkers and to screen out potential beneficial patients. Recent evidence has revealed that tumor microenvironment (TME) is highly associated with the prognosis of gastric cancer. Meanwhile, tumor microenvironment score (TMEscore) established with transcriptomic data is a robust biomarker for predicting prognosis and guiding individualized immunotherapy strategies. However, its predictive value for perioperative drug treatment outcomes warrants further exploration and validation. The study is a multi-center, observational study to evaluate the relationship between the efficacy of perioperative treatment and tumor microenvironment in patients with locally advanced resectable gastric and gastro-oesophageal junction adenocarcinoma, aiming at further determining the predictive value of TMEscore and establishing a comprehensive treatment-efficacy evaluation system for gastric cancer. Eligible subjects were selected according to the inclusion criteria and exclusion criteria. After the successful screening, the patients were treated in accordance with the clinical guidelines and the actual conditions. The residual tissue samples of the primary tumor were collected to conduct the tumor microenvironment detection. After routine neoadjuvant therapy, followed by a restaging of the tumor status and surgery. The residual surgical specimens were collected to conduct the tumor microenvironment detection analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced resectable gastric and gastro-oesophageal junction adenocarcinoma at the stage of cT2-T4aNxM0 (AJCC 8th) without distant metastases and without infiltration of adjacent structures and organs.
2. 18-75 years old.
3. Willing to provide residual tumor tissues after routine clinical diagnosis for tumor microenvironment detection analysis.
4. Patients agree to participate in the study and sign the informed consent.
5. Patients need to receive perioperative drug therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.

Exclusion Criteria:

1. Human epidermal growth factor receptor 2 (HER2) is positive, that is, tissue immunohistochemical staining (IHC) (3+) or IHC (2+), and tissue fluorescence in situ hybridization (FISH) is positive.
2. Patients with major cardiovascular and cerebrovascular diseases (such as congestive heart failure, unstable heart colic, atrial fibrillation, stroke, transient ischemic attack, etc.).
3. Allergies or contraindications to common chemotherapy drugs, immunotherapy drugs or the ingredients.
4. Women who are pregnant, breast-feeding.
5. Other conditions the investigator believes that it is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed locally advanced resectable gastric and gastro-oesophageal junction adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) rate | From the initiation date of first cycle to the date of surgery, an average of 10 weeks
  Defined as <10% residual viable tumor cells in the resection specimen after neoadjuvant drug treatment.

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate | From the initiation date of first cycle to the date of surgery, an average of 10 weeks
  Defined as the percentage of participants having a pathological complete response.
R0 resection rate | From the initiation date of first cycle to the date of surgery, an average of 10 weeks
  Rate of microscopically margin-negative resection.
Disease-free Survival (DFS) | 3 years
  Defined as the time from post-surgery baseline scan until the first occurrence of local/distant recurrence or death from any cause and is based on RECIST 1.1 as assessed by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No